CLINICAL TRIAL: NCT02750605
Title: Randomized Trial Comparing Drug Coated Balloon vs Plain Balloon Angioplasty in Critical Limb Ischemia and Treatment of Long Lesions in Crural Arteries
Brief Title: DEB ( Drug Eluting Balloon) in Crural Arteries and Critical Limb Ischemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Torbjorn Fransson, Consultant, Vascular Surgery, Skane University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TF3
Record Dates: First submitted 2016-01-19; First posted 2016-04-25 (Estimated); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Peripheral Vascular Diseases
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug eluting balloon angioplasty (Experimental): Intervention with DEB angioplasty in long lesions of crural arteries
  Interventions: Device: DEB
- Plain old balloon angioplasty (Active Comparator): Intervention with plain old balloon angioplasty POBA in long lesions of crural arteries
  Interventions: Device: POBA

INTERVENTIONS:
Device: DEB — Intervention with drug eluting balloon.
  Arms: Drug eluting balloon angioplasty
Device: POBA — Intervention with old technology as comparison
  Arms: Plain old balloon angioplasty

SUMMARY:
The purpose of this trial is to compare short- medium long-term results in treatment of PAD (peripheral arterial disease) in the crural arteries with either drug coated balloon or conventional balloons in a prospective , randomized, single center study

Results will be defined as:

Limb salvage, Event-free survival, Freedom from TLR (target lesion revascularization), Primary patency, Clinical success, Serious adverse events, and the patients will be followed-up for 1 years.

Primary endpoints:

Primary Patency at 12 months, TLR (clinical driven),

Secondary endpoints:

Event free survival, Clinical success at 6,12 months, Technical success, Serious adverse events,

ELIGIBILITY:
Inclusion Criteria:

* Critical limb ischemia. Rutherford class 4-6
* Crural disease, long lesions, more than 2 cm.
* Life expectancy > 1year
* > 18 years

Exclusion Criteria:

* Pregnancy
* Patients disapproval
* Allergy to drug or contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Primary patency of treated crural vessels | 12 months
  Evaluation with MRA (Magnetic Resonans Angiography) at 12 months, regarding binary restenosis or occlusion in the treated arterial segment. Proportion of treated segments that remains open.
Clinical driven target lesion revascularization (TLR) | 12 months
  Porportion of patients that needs retreatment in in the monitored arterial segment

CONTACTS AND LOCATIONS:
Overall Officials: Torbjörn Fransson, Principal Investigator — SUS, Malmö
Locations (1):
- Vascular center, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fransson T, Mohammed Y, Gottsater A, Resch T. Prospective Randomized Clinical Trial Comparing Paclitaxel-Coated Balloon Versus Conventional Balloon Angioplasty in Treating Below the Knee Arterial Lesions in Chronic Limb Threatening Ischemia: The CRURAL DEB Study. J Endovasc Ther. 2025 Nov 20:15266028251388746. doi: 10.1177/15266028251388746. Online ahead of print. PMID 41263159